CLINICAL TRIAL: NCT02877134
Title: A Phase 2b, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Multicenter Study to Evaluate the Safety and Efficacy of JnJ-64304500 in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: Safety and Efficacy Study of JNJ-64304500 in Participants With Moderately to Severely Active Crohn's Disease
Acronym: TRIDENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108136; 64304500CRD2001 (Other: Janssen Research & Development, LLC); 2016-000634-21 (EudraCT Number)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Results first posted 2022-02-17 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part I : Placebo (Experimental): Participants will receive placebo Subcutaneously (SC) at Weeks 0, 2, 4, 6, 8, and 10. From Week 12 Placebo-treated participants who are in clinical response at Week 12 (>=100-point reduction from baseline in Crohn's Disease Activity Index (CDAI) or CDAI <150) will continue to receive placebo SC injections every 2 weeks from Week 12 through Week 22. Placebo -treated participants who are not in clinical response at Week 12 will receive JNJ-64304500 400 mg SC at Week 12 and then JNJ-64304500 200 mg every two weeks from Week 14 through Week 22.
  Interventions: Drug: JNJ-64304500; Drug: Placebo
- Part I : JNJ-64304500 (Experimental): Participants will receive JNJ-64304500 400 milligram (mg) SC at Week 0 then 200 mg SC every two weeks through Week 22.
  Interventions: Drug: JNJ-64304500
- Part II : Placebo (Experimental): Placebo SC at Weeks 0, 2, 4, and 8. From Week 12, placebo-treated participants who are in clinical response at Week 12 (>=100-point reduction from baseline in CDAI or CDAI <150) will continue to receive placebo at Weeks 12, 14, 16, and 20. Placebo -treated participants who are not in clinical response at Week 12 will receive JNJ-64304500 150 mg SC at Week 12 and then JNJ-64304500 75 mg at Weeks 14, 16, and 20. Participants who complete Part II 24 weeks assessment and may benefit from continued treatment in the opinion of the investigator are eligible to enter the Part II LTE in which they will continue to receive placebo up to 52 weeks (for a total of up to 72 weeks of placebo in Part II).
  The study has been unblinded due to lack of sufficient efficacy of JNJ- 64304500. Participants receiving placebo during the LTE will stop receiving placebo.
  Interventions: Drug: JNJ-64304500; Drug: Placebo
- Part II : JNJ-64304500 High Dose (Experimental): JNJ-64304500 400 mg SC at Week 0 and 200 mg SC at Weeks 2, 4, 8, 12, 16, and 20. Participants who complete Part II 24 weeks assessment and may benefit from continued treatment in the opinion of the investigator are eligible to enter the Part II LTE in which they will continue to receive JNJ-64304500 high dose up to 52 weeks (for a total of up to 72 weeks of JNJ-64304500 in Part II).
  The study has been unblinded due to lack of sufficient efficacy of JNJ-64304500. Participants receiving JNJ-64304500 during the LTE will stop receiving study drug and will have a final safety follow-up visit 16 weeks after the last dose of study drug.
  Interventions: Drug: JNJ-64304500
- Part II : JNJ-64304500 Middle Dose (Experimental): JNJ-64304500 150 mg SC at Week 0 and 75 mg SC at Weeks 2, 4, 8, 12, 16, and 20. Participants who complete Part II 24 weeks assessment and may benefit from continued treatment in the opinion of the investigator are eligible to enter the Part II LTE in which they will continue to receive JNJ-64304500 middle dose up to 52 weeks (for a total of up to 72 weeks of JNJ-64304500 in Part II).
  The study has been unblinded due to lack of sufficient efficacy of JNJ-64304500. Participants receiving JNJ-64304500 during the LTE will stop receiving study drug and will have a final safety follow-up visit 16 weeks after the last dose of study drug.
  Interventions: Drug: JNJ-64304500
- Part II : JNJ-64304500 Low Dose (Experimental): JNJ-64304500 50 mg SC at Week 0 and 25 mg SC at Weeks 2, 4, 8, 12, 16, and 20. Participants who complete Part II 24 weeks assessment and may benefit from continued treatment in the opinion of the investigator are eligible to enter the Part II LTE in which they will continue to receive JNJ-64304500 low dose up to 52 weeks (for a total of up to 72 weeks of JNJ-64304500 in Part II).
  The study has been unblinded due to lack of sufficient efficacy of JNJ-64304500. Participants receiving JNJ-64304500 during the LTE will stop receiving study drug and will have a final safety follow-up visit 16 weeks after the last dose of study drug.
  Interventions: Drug: JNJ-64304500
- Part II : Ustekinumab (Experimental): Participants will receive tiered doses of Ustekinumab 260 mg (weight <=55 kg), Ustekinumab 390 mg (weight >55 kg and <=85 kg), Ustekinumab 520 mg (weight >85 kg) intravenously at Week 0 followed by 90 mg subcutaneously at Weeks 8 and 16. Participants who complete Part II 24 weeks assessment and may benefit from continued treatment in the opinion of the investigator are eligible to enter the Part II LTE in which they will continue to receive Ustekinumab up to 52 weeks (for a total of up to 72 weeks of Ustekinumab in Part II).
  The study has been unblinded due to lack of sufficient efficacy of JNJ-64304500. Participants receiving Ustekinumab during the LTE will stop receiving study drug and will have a final safety follow-up visit after the last dose of study drug. However, participants receiving Ustekinumab in countries where Ustekinumab is not commercially available or approved for adult Crohn's disease were continued to receive Ustekinumab in the LTE.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: JNJ-64304500 — Participants will receive JNJ-64304500 Subcutaneously.
  Arms: Part I : JNJ-64304500; Part I : Placebo; Part II : JNJ-64304500 High Dose; Part II : JNJ-64304500 Low Dose; Part II : JNJ-64304500 Middle Dose; Part II : Placebo
Drug: Placebo — Participants will receive placebo Subcutaneously.
  Arms: Part I : Placebo; Part II : Placebo
Drug: Ustekinumab — Participants will receive ustekinumab as per the dosing regimen.
  Other Names: STELARA
  Arms: Part II : Ustekinumab

SUMMARY:
The purpose of the study is to assess the safety and efficacy of JNJ-64304500 in participants with moderately to severely active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's disease or fistulizing Crohn's disease of at least 3 months' duration, with colitis, ileitis, or ileocolitis, confirmed at any time in the past by radiography, histology, and/or endoscopy
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [b-hCG]) pregnancy test result at screening and a negative urine pregnancy test result at Week 0
* Adhere to the following requirements for concomitant medication for the treatment of Crohn's disease, which are permitted provided that doses meeting these requirements are stable, or have been discontinued, for at least 3 weeks before baseline (Week 0), unless otherwise specified: a) Oral 5-aminosalicylic acid (5-ASA) compounds, b) Oral corticosteroids at a prednisone-equivalent dose at or below 40 milligram per day (mg/day), or 9 mg/day of budesonide, or 5 mg/day beclomethasone dipropionate, c) Antibiotics being used as a primary treatment of Crohn's disease, d) Conventional immunomodulators (that is, azathioprine (AZA), 6-mercaptopurine (6-MP), or Methotrexate (MTX)): participants must have been taking them for at least 12 weeks and at a stable dose for at least 4 weeks before baseline
* A participant who has had extensive colitis for greater than or equal to (>=) 8 years, or disease limited to the left side of the colon for >= 12 years, must either have had a colonoscopy to assess for the presence of dysplasia within 1 year before the first administration of study agent or a colonoscopy to assess for the presence of malignancy at the screening visit, with no evidence of malignancy
* Have active Crohn's disease, defined as a baseline Crohn's Disease Activity Index (CDAI) score of >= 220 but <= 450

Exclusion Criteria:

* Participants who have received intravenous (IV) corticosteroids less then (<)3 weeks or have received tumor necrosis factor-alpha (TNF-alpha) antagonist biologic agents (example, monoclonal antibody [mAb] therapies) or other agents intended to suppress or eliminate tumor necrosis factor-alpha (TNF-alpha) <8 weeks or have received Vedolizumab <16 weeks before the first administration of study drug
* Woman who is pregnant or planning pregnancy or is a man who plans to father while randomized in the study or within 16 weeks after the last administration of study agent
* Participants with certain complications of Crohn's disease that would make it hard to assess response to study drug
* Participants with a history of or ongoing chronic or recurrent infectious disease
* Has previously received a biologic agent targeting interleukin (IL)-12 or IL-23, including but not limited to ustekinumab or briakinumab (ABT-874)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (147):
- United States (37):
  - Lone Tree, Colorado
  - Coral Gables, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Miramar, Florida
  - Orlando, Florida
  - Winter Park, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Evanston, Illinois
  - Indianapolis, Indiana
  - Houma, Louisiana
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Columbia, Maryland
  - Morristown, New Jersey
  - Brooklyn, New York
  - Great Neck, New York
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Doylestown, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Southlake, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Richmond, Virginia
  - Seattle, Washington
- Belgium (3):
  - Brussels
  - Ghent
  - Liège
- Sofia, Bulgaria
- Canada (2):
  - Brandon, Manitoba
  - London, Ontario
- France (7):
  - Amiens
  - Lille
  - Marseille
  - Paris
  - Pierre-Bénite
  - Saint-Etienne
  - Toulouse
- Germany (11):
  - Berlin
  - Essen
  - Hamburg
  - Hanover
  - Heidelberg
  - Kiel
  - Leipzig
  - Ludwigshafen
  - Lübeck
  - Lüneburg
  - Ulm
- Hungary (4):
  - Budapest
  - Debrecen
  - Szekszárd
  - Szombathely
- Japan (30):
  - Asahikawa
  - Chikushino-shi
  - Fukushima
  - Gunma
  - Hamamatsu
  - Hirosaki
  - Hitachi
  - Hyôgo
  - Isehara
  - Kagoshima
  - Kahoku-gun
  - Kamakura
  - Kanagawa
  - Kanazawa
  - Kashiwa
  - Midori-ku
  - Minatoku
  - Niigata
  - Okinawa
  - Osaka
  - Ōsaka-sayama
  - Saga
  - Sakura
  - Sapporo
  - Sendai
  - Shimotsuga Gun
  - Shimotsuke
  - Shinjuku Ku
  - Shinjuku-ku
  - Sunto-gun
- Poland (12):
  - Bydgoszcz
  - Chorzów
  - Krakow
  - Ksawerów
  - Lodz
  - Oświęcim
  - Poznan
  - Sopot
  - Szczecin
  - Warsaw
  - Wroclaw
  - Włocławek
- Romania (3):
  - Bucharest
  - Oradea
  - Timișoara
- Russia (13):
  - Irkutsk
  - Kazan'
  - Krasnoyarsk
  - Moscov
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Tosno
  - Yekaterinburg
- South Korea (7):
  - Bundang
  - Busan
  - Daegu
  - Guri-si
  - Gyeonggi-do
  - Seoul
  - Suwon
- Ukraine (13):
  - Chernivtsi
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiyv
  - Kropyvnytskyi
  - Kyiv
  - Lviv
  - Sumy
  - Ternopil
  - Uzhhorod
  - Zaporizhzhia
  - Zhaporozhia
- United Kingdom (4):
  - Cambridge
  - Nottingham
  - Sheffield
  - Sutton in Ashfield

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993
- [Derived] Allez M, Sands BE, Feagan BG, D'Haens G, De Hertogh G, Randall CW, Zou B, Johanns J, O'Brien C, Curran M, Rebuck R, Wang ML, Sabins N, Baker T, Kobayashi T. A Phase 2b, Randomised, Double-blind, Placebo-controlled, Parallel-arm, Multicenter Study Evaluating the Safety and Efficacy of Tesnatilimab in Patients with Moderately to Severely Active Crohn's Disease. J Crohns Colitis. 2023 Aug 21;17(8):1235-1251. doi: 10.1093/ecco-jcc/jjad047. PMID 36939629

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In participant flow, data is reported in 2 periods, [Main Study" and "Part II long term extension (LTE) Phase"] depicts the information for the specified time period as: Part I: Through Week 38 (including safety follow-up); Part II: Through Week 24 for participants who entered the LTE phase and through Week 36 for participants who did not enter the LTE.
Groups:
- Part I: Placebo: Participants received placebo subcutaneously (SC) at Weeks 0, 2, 4, 6, 8, and 10. Participants in clinical response at Week 12 continued to receive placebo every 2 weeks (Q2W) through Week 22. Participants not in clinical response at Week 12 received JNJ-64304500 400 milligrams (mg) SC at Week 12 and then 200 mg SC Q2W from Week 14 through Week 22. Participants were followed up for safety up to Week 38.
- Part I: JNJ-64304500: Participants received JNJ-64304500 400 mg SC at Week 0 then 200 mg SC every two weeks through Week 22. All participants were followed up for safety up to Week 38.
- Part II: Placebo: Participants received placebo SC at Weeks 0, 2, 4, and 8. Participants in clinical response at Week 12 continued to receive placebo at Weeks 12, 14, 16, and 20. Participants not in clinical response at Week 12 received JNJ-64304500 150 mg SC at Week 12 and then JNJ-64304500 75 mg SC at Weeks 14, 16, and 20. Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II long term extension (LTE) phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II: JNJ-64304500 Low Dose: Participants received JNJ-64304500 50 mg SC at Week 0 and 25 mg SC at Weeks 2 and 4, then 25 mg SC every four weeks through Week 20. Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II LTE phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II: JNJ-64304500 Middle Dose: Participants received JNJ-64304500 150 mg SC at Week 0 and 75 mg SC at Weeks 2 and 4, then 75 mg SC every four weeks through Week 20. Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II LTE phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II: JNJ-64304500 High Dose: Participants received JNJ-64304500 400 mg SC at Week 0 and 200 mg SC at Weeks 2 and 4, then 200 mg SC every four weeks through Week 20. Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II LTE phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II: Ustekinumab: Participants received Ustekinumab (tiered doses approximating 6 milligrams/kilograms (mg/kg) intravenously [IV]) at Week 0 (as indicated in the bullets below), followed by 90 mg SC at Weeks 8 and 16. - Ustekinumab 260 mg (weight [less than or equal to [<=] 55 kg). - Ustekinumab 390 mg (weight greater than [>] 55 kg and less than or equal to [<=] 85 kg). Ustekinumab 520 mg (weight >85 kg). Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II LTE phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II LTE: Placebo: Participants randomized to placebo group and who were benefitted from continued treatment in the opinion of the investigator, entered the Part II LTE phase and received placebo or JNJ-64304500 middle dose (JNJ-64304500 75 mg SC) at Weeks 24, 28, 32, 36, 40, 44, 48, 52 56, 60, 64, 68, and 72. Participants were followed up for safety up to Week 88.
- Part II LTE: JNJ-64304500 Low Dose: Participants randomized to the 'JNJ-64304500 Low Dose' group and who were benefitted from continued treatment in the opinion of the investigator, entered the Part II LTE phase and received JNJ-64304500 25 mg SC at Weeks 24, 28, 32, 36, 40, 44, 48, 52 56, 60, 64, 68, and 72. Participants were followed up for safety up to Week 88.
- Part II LTE: JNJ-64304500 Middle Dose: Participants randomized to the 'JNJ-64304500 Middle Dose' group and who were benefitted from continued treatment in the opinion of the investigator, entered the Part II LTE phase and received JNJ-64304500 75 mg SC at Weeks 24, 28, 32, 36, 40, 44, 48, 52 56, 60, 64, 68, and 72. Participants were followed up for safety up to Week 88.
- Part II LTE: JNJ-64304500 High Dose: Participants randomized to the 'JNJ-64304500 High Dose' group and who were benefitted from continued treatment in the opinion of the investigator, entered the Part II LTE phase and received JNJ-64304500 200 mg SC at Weeks 24, 28, 32, 36, 40, 44, 48, 52 56, 60, 64, 68, and 72. Participants were followed up for safety up to Week 88.
- Part II LTE: Ustekinumab: Participants randomized to the 'Ustekinumab' group and who were benefitted from continued treatment in the opinion of the investigator, entered the Part II LTE phase and received Ustekinumab 90 mg IV at Weeks 24, 32, 40, 48, 56, 64 and 72. Participants were followed up for safety up to Week 88.
Period: Main Study (Parts I,II): Up to Week 38
Arm/Group | Part I: Placebo | Part I: JNJ-64304500 | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab | Part II LTE: Placebo | Part II LTE: JNJ-64304500 Low Dose | Part II LTE: JNJ-64304500 Middle Dose | Part II LTE: JNJ-64304500 High Dose | Part II LTE: Ustekinumab
Started | 72 | 73 | 48 | 50 | 49 | 49 | 47 | 0 | 0 | 0 | 0 | 0
Placebo Non Responders at Week 12 | 44 | 0 | 31 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 58 | 48 | 40 | 35 | 42 | 39 | 42 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 25 | 8 | 15 | 7 | 10 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 19 | 5 | 8 | 3 | 6 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 3 | 6 | 4 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Period: Part II LTE Phase: From Week 24-88
Arm/Group | Part I: Placebo | Part I: JNJ-64304500 | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab | Part II LTE: Placebo | Part II LTE: JNJ-64304500 Low Dose | Part II LTE: JNJ-64304500 Middle Dose | Part II LTE: JNJ-64304500 High Dose | Part II LTE: Ustekinumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 (Only eligible participants from main study phase, entered into Part II LTE phase.) | 21 (Only eligible participants from main study phase, entered into Part II LTE phase.) | 27 (Only eligible participants from main study phase, entered into Part II LTE phase.) | 24 (Only eligible participants from main study phase, entered into Part II LTE phase.) | 28 (Only eligible participants from main study phase, entered into Part II LTE phase.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 17 | 20 | 14 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 7 | 10 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 9 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I: Placebo | Part I: JNJ-64304500 | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab | Total
Number analyzed (Participants) | 72 | 73 | 48 | 50 | 49 | 49 | 47 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (13.3) | 38 (13.25) | 40.6 (13.69) | 36.4 (11.14) | 37.1 (15.04) | 37.2 (12.87) | 42 (12.62) | 38.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 24 | 16 | 27 | 20 | 23 | 174
  Male | 41 | 40 | 24 | 34 | 22 | 29 | 24 | 214
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 3 | 6 | 2 | 8 | 7 | 33
  Black or African American | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 67 | 63 | 45 | 43 | 46 | 39 | 40 | 343
  More than one race | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Other | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 4
  BULGARIA | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 7
  FRANCE | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
  GERMANY | 4 | 4 | 0 | 2 | 0 | 0 | 2 | 12
  HUNGARY | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  ITALY | 3 | 4 | 1 | 0 | 1 | 2 | 2 | 13
  JAPAN | 0 | 0 | 3 | 6 | 2 | 8 | 6 | 25
  POLAND | 14 | 9 | 5 | 7 | 17 | 11 | 9 | 72
  ROMANIA | 1 | 1 | 2 | 3 | 1 | 1 | 1 | 10
  RUSSIAN FEDERATION | 20 | 14 | 19 | 15 | 15 | 15 | 11 | 109
  SOUTH KOREA | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 6
  UKRAINE | 16 | 17 | 13 | 10 | 9 | 5 | 10 | 80
  UNITED KINGDOM | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 4
  UNITED STATES | 9 | 16 | 3 | 4 | 2 | 4 | 4 | 42

OUTCOME MEASURES:

1. Primary Outcome: Part I: Change From Baseline in the Crohn's Disease Activity Index (CDAI) Score at Week 8
Description: The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables. The CDAI score was assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s), and/or opiates, and general well-being. The last 4 variables were scored over 7 days by the participant on a diary card. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Time Frame: Baseline to Week 8
Population: The efficacy analyses were based on the Full analysis set (FAS) included all randomized participants in Part 1 who received at least 1 dose of study agent.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part I: Placebo | Part I: JNJ-64304500
Number analyzed (Participants) | 72 | 73
units on a scale | -60.0 (77.08) | -103.6 (93.54)

2. Primary Outcome: Part II: Change From Baseline in the CDAI Score at Week 12
Description: The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables. The CDAI was assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Time Frame: Baseline to Week 12
Population: FAS included all randomized participants in Part II who received at least 1 dose of study agent. Here 'N' refers to number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Part II: JNJ-64304500 Middle Dose: Participants received JNJ-64304500 150 mg SC at Week 0 and 75 mg SC at Weeks 2 and 4, then 75 mg SC every four weeks through Week 20. Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II long term LTE phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II: JNJ-64304500 High Dose: Participants received JNJ-64304500 400 mg SC at Week 0 and 200 mg SC at Weeks 2 and 4, then 200 mg SC every four weeks through Week 20. Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II long term LTE phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II: Ustekinumab: Participants received Ustekinumab (tiered doses approximating 6 milligrams/kilograms (mg/kg) intravenously [IV]) at Week 0 (as indicated in the bullets below), followed by 90 mg SC at Weeks 8 and 16. - Ustekinumab 260 mg (weight [less than or equal to [<=] 55 kg). - Ustekinumab 390 mg (weight greater than [>] 55 kg and less than or equal to [<=] 85 kg). Ustekinumab 520 mg (weight >85 kg). Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II long term LTE phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
Arm/Group | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab
Number analyzed (Participants) | 46 | 44 | 47 | 48 | 47
units on a scale | -59.2 (89.51) | -93.2 (117.91) | -72.2 (92.79) | -84.3 (103.28) | -148.8 (84.59)

3. Secondary Outcome: Part II: Percentage of Participants in Clinical Remission at Week 12 as Measured by CDAI (CDAI Less Than [<] 150)
Description: Clinical Remission was defined as a CDAI score of <150 point. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables. extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. A decrease in CDAI over time indicates improvement in disease activity. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Time Frame: Week 12
Population: FAS included all randomized participants in Part II who received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab
Number analyzed (Participants) | 48 | 50 | 49 | 49 | 47
percentage of participants | 14.6 | 30 | 18.4 | 22.4 | 53.2

4. Secondary Outcome: Part II: Percentage of Participants in Clinical Response at Week 12 as Measured by CDAI (Greater Than or Equal to [>=] 100-point Reduction From Baseline in CDAI or CDAI <150)
Description: Clinical response was defined as a >=100-point reduction from the baseline CDAI score, or a CDAI score <150. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables. extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Time Frame: Week 12
Population: FAS included all randomized participants in Part II who received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab
Number analyzed (Participants) | 48 | 50 | 49 | 49 | 47
percentage of participants | 22.9 | 42.0 | 40.8 | 30.6 | 72.3

5. Secondary Outcome: Part II: Change From Baseline in Patient-Reported Outcome (PRO)-2 at Week 12
Description: The PRO-2 score is defined as the sum of the abdominal pain and stool frequency components of the CDAI. PRO-2 scores ranges from 0 to approximately 300, higher score indicates higher disease activity.
Time Frame: Baseline, Week 12
Population: FAS included all randomized participants in Part II who received at least 1 dose of study agent. Here 'N' refers to the number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab
Number analyzed (Participants) | 46 | 44 | 47 | 48 | 46
units on scale | -28.8 (47.72) | -46.1 (59.14) | -39.8 (52.59) | -42.9 (47.33) | -70.1 (52.97)

6. Secondary Outcome: Part II: Percentage of Participants in Clinical Remission at Week 12 as Measured by PRO-2 (PRO-2 <75)
Description: Clinical Remission was defined as a PRO-2 score of <75 point.
Time Frame: Week 12
Population: FAS included all randomized participants in Part II who received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab
Number analyzed (Participants) | 48 | 50 | 49 | 49 | 47
percentage of participants | 16.7 | 32.0 | 30.6 | 44.9 | 53.2

7. Secondary Outcome: Part II: Percentage of Participants in Clinical Response at Week 12 as Measured by PRO-2 (>=50-point Reduction From Baseline in PRO-2 Score or PRO-2 Score <75)
Description: Clinical response was defined as >=50-point reduction from baseline in PRO-2 or Score or PRO-2 Score <75.
Time Frame: Week 12
Population: FAS included all randomized participants in Part II who received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab
Number analyzed (Participants) | 48 | 50 | 49 | 49 | 47
percentage of participants | 31.3 | 44.0 | 46.9 | 49.0 | 68.1

8. Secondary Outcome: Part II: Change From Baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 12
Description: SES-CD is a validated instrument reflecting an endoscopist global appraisal of mucosal lesions in Crohn's disease. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. The total SES-CD was calculated as the sum of the 4 variables for the 5 bowel segments: rectum, left colon, transverse colon, right colon, and ileum. Scores range from 0 to 60, with higher scores indicating more severe disease.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part II: Placebo | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab
Number analyzed (Participants) | 34 | 33 | 33 | 38 | 36
units on a scale | -2.2 (6.58) | -0.7 (6.47) | -1.2 (4.89) | -2.7 (6.93) | -2.6 (5.32)

ADVERSE EVENTS:
Time Frame: Part I: Through Week 38; Part II: Through Week 24 for participants who entered the LTE and through Week 36 for participants who did not enter the LTE; Part II LTE: from Week 24 through Week 88
Description: The Safety Analysis Set included all randomized participants who received at least 1 dose of study agent (placebo or JNJ-64304500 or ustekinumab, including a partial dose).
Groups:
- Part I: Placebo: Participants received placebo subcutaneously (SC) at Weeks 0, 2, 4, 6, 8, and 10. Participants in clinical response at Week 12 continued to receive placebo every 2 weeks (Q2W) through Week 22. Participants not in clinical response at Week 12 received JNJ-64304500 400 mg SC at Week 12 and then 200 mg SC Q2W from Week 14 through Week 22. Safety results included data up to the time of receiving JNJ-64304500 for those who received JNJ-64304500 at Week 12 and included all data for those who did not receive JNJ-64304500 at Week 12. Participants were followed up for safety up to Week 38.
- Part I: Placebo to JNJ-64304500: Participants received placebo SC at Weeks 0, 2, 4, 6, 8, and 10. Participants in clinical response at Week 12 continued to receive placebo Q2W through Week 22. Participants not in clinical response at Week 12 received JNJ-64304500 400 mg SC at Week 12 and then 200 mg SC Q2W from Week 14 through Week 22. Safety results included data from the time of receiving JNJ- 64304500 at Week 12 onward. Participants were followed up for safety up to Week 38.
- Part I: JNJ-64304500: Participants received JNJ-64304500 400 mg SC at Week 0 then 200 mg SC every two weeks through Week 22. Participants were followed up for safety up to Week 38.
- Part II: Placebo: Participants received placebo SC at Weeks 0, 2, 4, and 8. Participants in clinical response at Week 12 continued to receive placebo at Weeks 12, 14, 16, and 20. Participants not in clinical response at Week 12 received JNJ 64304500 150 mg SC at Week 12 and then JNJ-64304500 75 mg SC at Weeks 14, 16, and 20. Safety results included data up to the time of receiving JNJ- 64304500 for those who received JNJ-64304500 at Week 12 and included all data for those who did not receive JNJ-64304500 at Week 12. Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II long term extension (LTE) phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II: Placebo to JNJ-64304500 Middle Dose: Participants received placebo SC at Weeks 0, 2, 4, and 8. Participants in clinical response at Week 12 continued to receive placebo at Weeks 12, 14, 16, and 20. Participants not in clinical response at Week 12 received JNJ 64304500 150 mg SC at Week 12 and then JNJ-64304500 75 mg SC at Weeks 14, 16, and 20. Safety results included data from the time of receiving JNJ- 64304500 at Week 12 onward. Participants who completed Part II Week 24 assessments and who were benefited from continued treatment, in the opinion of the investigator, were eligible to enter the Part II LTE phase at Week 24. Participants who did not enter into LTE phase at Week 24 were followed up for safety up to Week 36.
- Part II LTE: Placebo: Participants randomized to placebo group and who were benefitted from continued treatment in the opinion of the investigator, entered the Part II LTE phase and received placebo at Weeks 24, 28, 32, 36, 40, 44, 48, 52 56, 60, 64, 68, and 72. Participants were followed up for safety up to Week 88.
- Part II LTE: Placebo to JNJ-64304500 Middle Dose: Participants randomized to placebo group and had dose adjustment to JNJ-64304500 middle dose at Week 12 and continued to receive JNJ-64304500 middle dose (JNJ-64304500 75 mg) SC at Weeks 24, 28, 32, 36, 40, 44, 48, 52 56, 60, 64, 68, and 72 in the Part II LTE. Participants were followed up for safety up to Week 88.
Arm/Group | Part I: Placebo | Part I: Placebo to JNJ-64304500 | Part I: JNJ-64304500 | Part II: Placebo | Part II: Placebo to JNJ-64304500 Middle Dose | Part II: JNJ-64304500 Low Dose | Part II: JNJ-64304500 Middle Dose | Part II: JNJ-64304500 High Dose | Part II: Ustekinumab | Part II LTE: Placebo | Part II LTE: Placebo to JNJ-64304500 Middle Dose | Part II LTE: JNJ-64304500 Low Dose | Part II LTE: JNJ-64304500 Middle Dose | Part II LTE: JNJ-64304500 High Dose | Part II LTE: Ustekinumab
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/44 | 1/73 | 0/48 | 0/31 | 0/50 | 0/49 | 1/49 | 0/47 | 0/10 | 0/12 | 0/21 | 0/27 | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/72 | 2/44 | 8/73 | 3/48 | 0/31 | 3/50 | 0/49 | 6/49 | 2/47 | 1/10 | 3/12 | 2/21 | 5/27 | 5/24 | 5/28
Other Adverse Events (participants affected / at risk) | 24/72 | 10/44 | 38/73 | 16/48 | 6/31 | 24/50 | 23/49 | 26/49 | 20/47 | 5/10 | 5/12 | 6/21 | 12/27 | 10/24 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Placebo (N=72) | Part I: Placebo to JNJ-64304500 (N=44) | Part I: JNJ-64304500 (N=73) | Part II: Placebo (N=48) | Part II: Placebo to JNJ-64304500 Middle Dose (N=31) | Part II: JNJ-64304500 Low Dose (N=50) | Part II: JNJ-64304500 Middle Dose (N=49) | Part II: JNJ-64304500 High Dose (N=49) | Part II: Ustekinumab (N=47) | Part II LTE: Placebo (N=10) | Part II LTE: Placebo to JNJ-64304500 Middle Dose (N=12) | Part II LTE: JNJ-64304500 Low Dose (N=21) | Part II LTE: JNJ-64304500 Middle Dose (N=27) | Part II LTE: JNJ-64304500 High Dose (N=24) | Part II LTE: Ustekinumab (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 1 | 5 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 4 | 0 | 1
Ileal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Device Related Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Placebo (N=72) | Part I: Placebo to JNJ-64304500 (N=44) | Part I: JNJ-64304500 (N=73) | Part II: Placebo (N=48) | Part II: Placebo to JNJ-64304500 Middle Dose (N=31) | Part II: JNJ-64304500 Low Dose (N=50) | Part II: JNJ-64304500 Middle Dose (N=49) | Part II: JNJ-64304500 High Dose (N=49) | Part II: Ustekinumab (N=47) | Part II LTE: Placebo (N=10) | Part II LTE: Placebo to JNJ-64304500 Middle Dose (N=12) | Part II LTE: JNJ-64304500 Low Dose (N=21) | Part II LTE: JNJ-64304500 Middle Dose (N=27) | Part II LTE: JNJ-64304500 High Dose (N=24) | Part II LTE: Ustekinumab (N=28)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 9 | 3 | 0 | 6 | 7 | 2 | 1 | 0 | 1 | 0 | 3 | 1 | 2
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 3 | 5 | 1 | 1 | 2 | 1 | 3 | 5 | 1 | 0 | 1 | 0 | 0 | 2
Crohn's Disease (Gastrointestinal disorders) | 4 | 0 | 6 | 4 | 0 | 4 | 7 | 2 | 2 | 1 | 1 | 1 | 4 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Enterovesical Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 3 | 3 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 1 | 1 | 4 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 7 | 2 | 1 | 3 | 3 | 4 | 4 | 0 | 1 | 1 | 3 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 2 | 0 | 7 | 1 | 0 | 2 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Platelet Count Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Tumour Inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 8 | 3 | 0 | 2 | 4 | 4 | 5 | 1 | 1 | 0 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT02877134/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT02877134/SAP_001.pdf